CLINICAL TRIAL: NCT01410539
Title: Mechanism Of Stent Thrombosis (MOST) Study, a Prospective Multicentre Non-randomized Registry
Brief Title: Mechanism Of Stent Thrombosis (MOST) Study
Acronym: Most
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, David Antoniucci, Head Division of Invasive Cardiology, Careggi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOST Study
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Artery; Stent Thrombosis; Platelet; Thrombus
Keywords: Stent Thrombosis; Percutaneous Coronary Intervention; Bare Metal Stent; Drug Eluting Stent; Residual Platelet Reactivity; Optical Coherence Tomography; OCT
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent Thrombosis (Experimental): Consecutive patients with stent thrombosis with stent strut assessment by OCT
  Interventions: Device: OCT guided PCI
- Controls (Active Comparator): Control subjects without stent thrombosis from the RHR OCT database
  Interventions: Drug: OCT guided medical therapy

INTERVENTIONS:
Device: OCT guided PCI — OCT guided PCI. Only thrombectomy in case of negative OCT findings (other than uncovered struts).
  Arms: Stent Thrombosis
Drug: OCT guided medical therapy — OCT guided medical therapy. Tailored antiplatelet therapy.
  Arms: Controls

SUMMARY:
This study is designed to assess the pathophysiology of ST by studying the main procedural and anatomical factors involved in the genesis of ST such as those related to stent and the vascular wall, as well as to the individual platelet residual reactivity.

ELIGIBILITY:
Inclusion Criteria:

* previous PCI with bare metal stent (BMS) or drug eluting stent (DES) and a definite subacute coronary ST
* previous PCI with DES and a definite late or very late coronary ST

Exclusion Criteria:

* Development of ST within 72 hours of stent implantation (acute and early subacute ST).
* Late and very late ST of BMS.
* Absence of informed consent.
* Age less than 18 years.
* Creatinine values greater than 2.5 g/dl (this is to avoid the negative effects related to the contrast medium necessary to perform the OCT evaluation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Percentage of uncovered stent struts | After thrombectomy
  The percentage of uncovered stent struts by OCT in patients with subacute stent thrombosis (either DES and BMS) and the percentage of uncovered stent struts in patients with late (after one month) and very late thrombosis of DES.

SECONDARY OUTCOMES:
Percentage of malapposed stent struts | After Thrombectomy
  The percentage of malapposed stent struts by OCT in patients with subacute thrombosis of DES and BMS and the percentage of malapposed stent struts by OCT in patients with late and very late thrombosis of DES.
Percentage of patients with high residual platelet reactivity | Baseline
  The percentage of patients with residual platelet reactivity (RPR) to ADP and arachidonic acid identified by values ≥ 240 P2Y12 reaction units (PRU) and ≥ 550 aspirin reaction units (ARU), respectively,. during aspirin and clopidogrel therapy or in which one or both the antiplatelet drugs have been interrupted.

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Study Chair — Careggi Hospital, Division of Invasive Cardiology; Francesco Prati, MD, Principal Investigator — Rome Heart Research
Locations (1):
- Careggi Hospital, Department of Hearth and Vessels, Florence, Italy

REFERENCES:
- [Derived] Parodi G, La Manna A, Di Vito L, Valgimigli M, Fineschi M, Bellandi B, Niccoli G, Giusti B, Valenti R, Cremonesi A, Biondi-Zoccai G, Prati F. Stent-related defects in patients presenting with stent thrombosis: differences at optical coherence tomography between subacute and late/very late thrombosis in the Mechanism Of Stent Thrombosis (MOST) study. EuroIntervention. 2013 Dec;9(8):936-44. doi: 10.4244/EIJV9I8A157. PMID 24384290